CLINICAL TRIAL: NCT03730675
Title: Irradiation Stent Placement Plus Transcatheter Arterial Chemoembolization in Hepatocellular Carcinoma With Portal Vein Tumor Thrombosis: A Multicenter Randomized Study
Brief Title: Irradiation Stent Placement Plus TACE for HCC and PVTT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, President, Zhongda Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZhongdaH-PATENCY
Record Dates: First submitted 2018-10-28; First posted 2018-11-05 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Hepatocellular Carcinoma; Portal Vein Tumor Thrombosis
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- irradiation stent plus TACE (Experimental): Portal irradiation stent placement will be performed before TACE procedures.
  Interventions: Procedure: Portal irradiation stent placement; Procedure: TACE
- Sorafenib plus TACE (Active Comparator): TACE will be performed in patients randomized to Arm B, with sequential sorafenib.
  Interventions: Procedure: TACE; Drug: Sorafenib

INTERVENTIONS:
Procedure: Portal irradiation stent placement — The irradiation portal vein stent was designed as two separate parts that consisted of an outer seeds-loaded-stent and an inner self-expandable metallic stent
  Arms: irradiation stent plus TACE
Procedure: TACE — TACE is a minimally invasive procedure performed in interventional radiology to restrict a tumor's blood supply.
Drug: Sorafenib — Sorafenib is a kinase inhibitor drug approved for the treatment of advanced hepatocellular carcinoma.
  Arms: Sorafenib plus TACE

SUMMARY:
The study is a multicenter, randomized (1:1), open-label, parallel-arm, Phase 3 clinical trial to evaluate the efficacy and safety of portal irradiation stent placement plus TACE compared to sorafenib plus TACE in patients with advanced HCC accompanied by portal vein tumor thrombosis. Patients will be randomized to receive either portal irradiation stent placement plus TACE(Arm A) or Sorafenib plus TACE (Arm B).

DETAILED DESCRIPTION:
The prognosis of HCC with portal vein tumor thrombosis (PVTT) is dismal, with a median survival of 2.7-4.0 months compared to that of 10.0-24.0 months without PVTT. Therefore, the presence of PVTT is regarded as a hallmark of advanced HCC and has a high incidence of 39-63%.

PVTT can accompany intrahepatic tumor spread, liver function deterioration, and portal vein hypertension, and can lead to intractable ascites, variceal rupture, hepatic encephalopathy and/or death. As recommended by the Barcelona Clinic Liver Cancer (BCLC) group, the current standard treatment of HCC with PVTT is sorafenib only. However, sorafenib monotherapy does not achieve satisfactory outcomes, yielding a median survival time of 5.6 to 8.1 months. To improve the prognosis, transarterial chemoembolization (TACE), surgical resection, radiotherapy, ablations, and radioembolization have been applied to treat patients with HCC and PVTT, with improved outcomes reported.

Portal vein stent placement is regarded as a safe and effective technique in relieving portal hypertension, extending treatment options, and prolonging survival in patients with HCC and PVTT. However, the reported stent patency period of 3.7 months and survival time of 2.2 to 6.1 months may not be interpreted as satisfactory outcomes, mainly limited by rapid tumor infiltration and/or subsequent thrombosis formation.

An irradiation stent has been developed and confirmed to be safe and effective in treating unresectable esophageal cancer. A modified irradiation stent designed for biliary tract obstruction was subsequently developed and resulted in significantly improved outcomes in a single-institute randomized, controlled study of patients with malignant biliary obstruction. This study aims to demonstrate that overall survival on portal irradiation stent placement plus TACE is superior to overall survival on sorafenib plus TACE in patients with advanced hepatocellular carcinoma accompanied by portal vein tumor thrombosis. Secondary Objectives includes 1. To compare time to progression between both treatment groups; 2. To compare hepatic function between both treatment groups; 3.To compare the disease control rate of the intrahepatic lesions between both treatment groups; 4.To evaluate and compare the safety and tolerability of both treatment groups; 5. To compare portal patency both treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* •

  1. Histologically-confirmed or clinical diagnosis of hepatocellular carcinoma (HCC)
  2. Histologically-confirmed or imaging-based diagnosis malignant portal vein tumor thrombosis(PVTT)
  3. Portal trunk invaded tumor thrombosis without the infiltration of superior mesenteric vein or inferior caval vein
  4. At least one patent first branch of the portal vein
  5. Measurable intrahepatic disease according to mRECIST
  6. Child-Pugh class A or B
  7. Eighteen years of age or older
  8. With an expected lifespan more than 3 months
  9. ECOG performance status 0, 1 or 2
  10. Required baseline laboratory data within the following parameters:

  1. Neutrophils ≥ 1.0×10⁹/L 2. Platelets ≥ 50×10⁹ /L 3. Hemoglobin ≥ 90 g/L 4. Serum aspartate aminotransferase (AST; ALT≤5 x ULN) 5. Serum creatinine ≤1.5 x ULN 6. INR <1.7 or prothrombin time (PT) < 4 seconds above ULN 7. Total bilirubin < 34.2 umol/L(2 mg/dL) 11. Signed and dated informed consent and willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures

Exclusion Criteria:

1. Presence of distant metastasis outside liver or diagnosis of any second malignancy beyond HCC
2. Less than 30% volume of uninvolved liver
3. Prior systemic treatment, including prior treatment with sorafenib or any prior local therapy (such as surgery, radiation therapy, hepatic arterial embolization, TACE, hepatic arterial infusion, radiofrequency ablation, percutaneous ethanol injection or cry ablation)
4. Presence of clinically relevant ascites (that can be classified as Child-Pugh score of 3).
5. Documented variceal hemorrhage within 6 months of study entry or presence of esophageal varices at risk of bleeding (as documented by endoscopy/CT/fluoroscopy)
6. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of study entry
7. Any of the following within the 3 months prior to study drug administration: severe/unstable angina, myocardial infarction, coronary artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, including transient ischemic attack, or pulmonary embolism.
8. Ongoing cardiac dysrhythmias of NCI CTCAE grade≥2, atrial fibrillation of any grade, or prolongation of the QTc interval to > 450 msec for males or > 470 msec for females.
9. Hypertension that cannot be controlled by medications (blood pressure >150/100 mm Hg despite optimal medical therapy).
10. Concomitant treatment with botanical formulation having an approved indication for cancer treatment, such as "Xiao Chai Hu Tang", "Kanglaite", "Huai Er Ke Li"etc.
11. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
12. Pregnancy or breastfeeding. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) within the 7 days prior to study enrollment.
13. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2018-11-10 (Actual); Primary Completion 2021-11-10 (Estimated); Study Completion 2021-11-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival | up to 36 months
  Overall survival was measured from the date of randomization until the date of death from any cause.

SECONDARY OUTCOMES:
Hepatic function in terms of albumin and total bilirubin | up to 36 months
  Hepatic function was measured in terms of albumin and total bilirubin.
Time to symptomatic progression | up to 36 months
  The time to symptomatic progression was measured from the date of randomization until the first documented event of symptomatic progression. Symptomatic progression was defined as a deterioration in ECOG performance status to 4 or death
Patency of portal vein | up to 36 months
  Patency of portal vein was evaluated by color doppler ultrasound
Disease control rate of intrahepatic lesions | up to 36 months
  Disease control rate of intrahepatic lesions referred to percentage of patients who had complete response, partial response, or stable disease.
Treatment Safety in terms of type, incidence, severity timing, seriousness, and relatedness of adverse events and laboratory abnormalities | up to 36 months
  Safety was evaluated in terms of type, incidence, severity (graded by the Common Terminology Criteria for Adverse Events [CTCAE], version 4.02), timing, seriousness, and relatedness of adverse events and laboratory abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, M.D., Principal Investigator — Zhongda Hospital
Locations (1):
- Zhong-da Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lu J, Guo JH, Ji JS, Li YL, Lv WF, Zhu HD, Sun JH, Ren WX, Zhang FJ, Wang WD, Shao HB, Cao GS, Li HL, Gao K, Yang P, Yin GW, Zhu GY, Wu FZ, Wang WJ, Lu D, Chen SQ, Min J, Zhao Y, Li R, Lu LG, Lau WY, Teng GJ. Irradiation stent with 125 I plus TACE versus sorafenib plus TACE for hepatocellular carcinoma with major portal vein tumor thrombosis: a multicenter randomized trial. Int J Surg. 2023 May 1;109(5):1188-1198. doi: 10.1097/JS9.0000000000000295. PMID 37038986